CLINICAL TRIAL: NCT04683094
Title: Comparative Study for the Validity of Various Severity Scoring System in the Surgical Intensive Care Unit at Aswan University Hospital
Brief Title: Comparative Study for the Validity of Various Severity Scoring System
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Huda Fahmy Mahmoud, PhD, Assistant professor of Anesthesia and Intensive Care, Aswan University Hospital
Other Study IDs: 449/3/20
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Head Trauma; Polytrauma; Pre-Eclampsia; Sepsis; Septic Shock
Keywords: APACH IV; SAPS III , SOFA score
MeSH Terms: conditions — Craniocerebral Trauma; Multiple Trauma; Pre-Eclampsia; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scoring systems for use in intensive care unit (ICU) patients have been introduced and developed over the last 30 years. They allow an assessment of the severity of disease and provide an estimate of in-hospital mortality

DETAILED DESCRIPTION:
Severity scoring systems that are commonly used in critical care settings include Acute Physiology and Chronic Health Evaluation (APACHE), which was developed in the 1980s for predicting mortality, Simplified Acute Physiology Score (SAPS), and Mortality Probability Model (MPM). Although these scoring systems use different variables and weights for the classification of disease severity, they commonly monitor parameters such as heart rate, blood pressure, neurological state, and clinical data as these factors significantly deviate from physiological normality in the progression of critical disease. Old age and chronic disease are also captured by the scoring systems. Sequential Organ Failure Assessment (SOFA) score, which is based on organ failure over time to evaluate morbidity and multiple organ dysfunction is also used.

ELIGIBILITY:
Inclusion Criteria:

* newly admitted patients to the Surgical Intensive Care Unit with head trauma multiple trauma craniotomy sepsis preeclampsia - eclampsia postop. for vascular surgery

Exclusion Criteria:

less than 16 years old, readmitted to the ICU during the study period as only the first admission will be considered, ICU length of stay (LOS) less than 24 h

Ages: 16 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: newly admitted patients to the Surgical Intensive Care Unit at Aswan University Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation (APACHE) IV | the first 24 hours after ICU admission
Simplified Acute Physiology Score (SAPS III) | the first 24 hours after ICU admission
Sequential Organ Failure Assessment (SOFA) score | the first 24 hours after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: huda fahmy, Principal Investigator — Aswan University
Locations (1):
- Huda Fahmy, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided